CLINICAL TRIAL: NCT05718323
Title: A Single-arm Phase II Trial of the Addition of Niraparib to Anti-PD-L1 Antibody Maintenance in Patients With SLFN11-positive, Extensive-disease Small Cell Lung Cancer.
Brief Title: Niraparib Added to Anti-PD-L1 Antibody Maintenance in SLFN11-positive, Extensive-disease SCLC
Acronym: RAISE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: GlaxoSmithKline (Industry); Development Limited (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 23-22
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: SCLC,Extensive Stage; SLFN11-positive
MeSH Terms: interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — 200 mg orally once daily, until PD 300 mg once daily if body weight ≥77 kg and platelets ≥150 g/L, until PD

SUMMARY:
RAISE is an international, multicentre, single-arm phase II trial. The trial treatment consists of the addition of niraparib, 200 mg orally once daily to anti-PD-L1 antibody maintenance. The primary objective of this trial is to assess the clinical efficacy of the addition of niraparib to anti-PD-L1 monoclonal antibody maintenance treatment in patients with SLFN11-positive ED-SCLC which has not progressed following standard first-line chemo-immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for SLFN11-expression testing

* Written IC part 1: for SLFN11-screening must be signed and dated by the patient and the investigator prior to sending any tumour material to the central laboratory.
* Histologically or cytologically confirmed ED-SCLC (stage IV according to the 8th TNM classification).
* Availability of FFPE tumour tissue for screening.

Inclusion criteria for trial participation

* Written IC part 2: for trial participation must be signed and dated by the patient and the investigator prior to any trial-related intervention.
* High SLFN11-expression on FFPE tumour material:

SLFN11-expression is determined at the central screening laboratory in Basel. Overexpression is defined as detectable protein expression by IHC in ≥20% of tumour cells.

* Patients must have received standard first-line chemo-immunotherapy, consisting of 4 cycles of platinum-etoposide chemotherapy in combination with an anti-PD-L1 antibody (atezolizumab or durvalumab). Patients who started the immunotherapy at chemotherapy cycle 2 are eligible.
* ED-SCLC must not have progressed during or after standard chemo-immunotherapy (as per RECIST v1.1).
* Patients must be candidates for ongoing maintenance treatment with immune-checkpoint inhibition.
* Adequate haematological function:
* Adequate renal function:
* Adequate liver function:
* ECOG PS 0-2
* Age ≥18 years
* Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum pregnancy test within 4 weeks before enrolment and within 3 days before treatment start.

Exclusion Criteria:

* Symptomatic brain metastases
* Any clinically active cancer, other than SCLC Exception: malignancies with negligible risk of metastases or death (e.g. 5-year OS rate of >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localised prostate cancer, ductal carcinoma in situ, or stage I uterine cancer. Hormonal therapy for non-metastatic prostate or ductal carcinoma in situ is allowed.

Consolidating thoracic radiotherapy. Palliative radiotherapy to the brain or to bones is allowed.

* History of idiopathic pulmonary fibrosis, organising pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
* Any lung disease requiring systemic steroids in doses of >10 mg prednisolone (or equivalent dose of other steroid).
* Any serious concomitant systemic disorders (for example active infection, unstable cardiovascular disease) which in the opinion of the investigator would compromise the patient's ability to complete the trial or interfere with the evaluation of the efficacy and safety of the protocol treatment.
* Inadequately controlled hypertension, defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >95 mmHg.

The patient must be considered stable and hypertension medically controlled.

* History of myelodysplastic syndrome/acute myeloid leukemia (MDS/AML).
* Prior Reversible Encephalopathy Syndrome (PRES)
* Severe renal or hepatic impairment.
* Any clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels.
* Treated with live vaccine within 30 days before enrolment.
* Hypersensitivity to niraparib or any of its excipients (e.g., tartrazine).
* Women who are pregnant or in the period of lactation.
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the trial and within the required timelines after last dose of niraparib treatment.
* Judgment by the investigator that the patient is unlikely to comply with trial procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 3 months by investigator assessment (according to RECIST v1.1) | From date of enrolment until 3 months post-enrolment
  Defined as the rate of patients without a PFS event at 3 months after enrolment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the date of enrolment until last tumour assessment (approximately 25-30 months after the enrolment of the first patient)
  Defined as the time from the date of enrolment until documented progression
Overall survival (OS) | From the date of enrolment until death from any cause (approximately 25-30 months after the enrolment of the first patient)
  Defined as the time from the date of enrolment until death from any cause
Disease control rate (DCR) by investigator assessment (according to RECIST v1.1) | approximately 25-30 months after the enrolment of the first patient
  Defined as the rate of patients, among all enrolled patients, that achieve a complete response (CR) or partial response (PR) or stabilisation of disease (SD, at least at week 6) by investigator assessment
Adverse events according to CTCAE v5.0 | From the date of enrolment until last patient last visit (approximately 25- 30 months after enrolment of the first patient)
  Adverse events according to CTCAE v5.0 (any-cause as well as treatment-related) including adverse events leading to dose interruptions, withdrawal of protocol treatment and death

CONTACTS AND LOCATIONS:
Overall Officials: Markus Joerger, MD-PhD, Study Chair — Department of Medical Oncology, Cantonal Hospital St.Gallen
Locations (18):
- France (4):
  - CHU - Angers, Angers
  - Centre Hospitalier d'Avignon, Avignon
  - Caen - CHU, Caen
  - Lyon - Centre Léon Bérard, Lyon
- Italy (4):
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola
  - Instituto Europeo di Oncologia (IEO), Milan
  - Santa Maria della Misericordia Hospital, Perugia
  - AULSS2 Marca Trevigiana Treviso, Treviso
- Spain (3):
  - Complejo Hospitalario Universitario a Coruña, A Coruña
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Puerta de Hierro, Madrid
- Switzerland (7):
  - Kantonsspital Baden, Baden
  - University Hospital Basel, Basel
  - Inselspital Bern, Bern
  - Kantonsspital St. Gallen, Sankt Gallen
  - Centre Hospitalier du Valais Romand, Sion
  - Bürgerspital Solothurn, Solothurn
  - Kantonsspital Winterthur, Winterthur

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP